CLINICAL TRIAL: NCT02166307
Title: Clinical Verification of Peptide Biomarkers for Human Aging by Standard-Free, Label-Free LC-MS/MS Quanification of Aldehyde-modified Peptides
Brief Title: Clinical Verification of Peptide Biomarkers for Human Aging
Status: Completed | Type: Observational
Sponsor: Beijing Institute of Technology (Other)
Responsible Party: Principal Investigator, Yulin Deng, Dean of School of Life Science, Beijing Institute of Technology
Other Study IDs: deng02
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Aging
Keywords: formaldehyde; Maillard Reaction; cross-linkage; human aging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aging in human physically refers to a multidimensional process that all the changes were accumulated in a person over time. These aging changes are responsible for the progressive increases in the chance of disease and death associated with them. So far, there are several theories have been developed to understand the aging process, such as cross-linking, which is led by Maillard Reactions. Maillard Reaction is a complex series of reactions between reducing sugar/aldehydes and amino groups on proteins. Under physiological conditions, aldehydes are products of various exogenous and endogenous amines catalyzed by semicarbazide-sensitive amine oxidase (SSAO), a family of heterogeneous enzyme. It was reported that SSAO shows a significant higher catalytic activity, producing more aldehydes in age-related diseases. However, SSAO is not a perfect candidate to be monitored for evaluating aging, because it is widely distributed in tissues, which are not readily accessible sample-sources for clinical applications. In this work, the investigators have found 6 biomarker candidates by developing a standard-free, label-free MS-based proteomics method based on standard protein (human serum albumin, the highest abundance protein in human plasma) model in vitro. Then, the investigators wanted to verify these biomarker candidates by clinical plasma samples to see if there is significant quantitative difference among people with different ages.

DETAILED DESCRIPTION:
The procedure of clinical study was:

1. to get plasma samples from hospital;
2. digestion of plasma protein-mixture by trypsin in lab;
3. run mass spectrometry and monitor the amount of target HSA-peptides.

ELIGIBILITY:
Inclusion Criteria:

* Cases with different ages

Exclusion Criteria:

* Cases with Diabetes Mellitus and Hepatitis B

Ages: 23 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: university hospital, plasma samples of physical examination, faculties and staff of a certain university
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
measurement of the amount of plasma peptides | two years
  The investigators have found 6 biomarker candidates by developing a standard-free, label-free MS-based proteomics method based on standard protein (human serum albumin, the highest abundance protein in human plasma) model in vitro. Then, the investigators wanted to verify these biomarker candidates by clinical plasma samples to see if there is significant quantitative difference among people with different ages.

CONTACTS AND LOCATIONS:
Overall Officials: Yulin Deng, Ph.D, Principal Investigator — School of Life Science, BIT